CLINICAL TRIAL: NCT05616663
Title: SARS-COV-2 Infection Among Hospital Staff: Study of Professional and Individual Factors of Covi-19 and Impact on Return to Work
Brief Title: Study of Professional and Individual Factors of Covi-19 and Impact on Return to Work
Acronym: FP-COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7954
Record Dates: First submitted 2022-11-14; First posted 2022-11-15 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Started on January 9, 2020 with the announcement of the discovery of a new SARS-CoV-2 coronavirus, the Covid-19 pandemic is responsible as of June 21, 2020 for 160,377 confirmed cases in France, 29,640 deaths and 9,823 hospitalizations. The Grand Est region is one of the regions in France that was most precociously and strongly affected by the epidemic, in particular the Strasbourg University Hospital. Faced with the heavy use of the healthcare system, hospital staff of all categories are an essential resource to be preserved. Several studies have shown the significant impact of Covid-19 on doctors and caregivers. In order to better protect these personnel and avoid contamination that could be harmful to their health but also because of the consequences in terms of staff, it is necessary to better understand the risk factors for transmission of this infection, the means of protection, the evolution of the disease and the determinants of the return to work. Few studies have explored on such a large workforce and in detail the professional risk factors for developing Covid-19 within different groups of hospital professionals including also non-caregivers and the evolution when returning to work in an outpatient population.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Professionals from the University Hospitals of Strasbourg (HUS)
* Professionals who had been working at the HUS at the time of the diagnosis of SARS CoV-2 infection.
* Subject having not expressed, after being informed, opposition to the reuse of their data for research purposes

Exclusion criteria:

- Subject who expressed their opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Professional rom the University Hospitals of Strasbourg (HUS) who had been working at the HUS at the time of the diagnosis of SARS CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 639 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-12-16 (Estimated); Study Completion 2023-12-16 (Estimated)

PRIMARY OUTCOMES:
positive RT-PCR test | one week after infection with Covid-19
  The presence of SARS CoV 2 infection is assessed by a positive RT-PCR test

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pathologie Professionnelle et Médecine du Travail - CHU de Strasbourg - France, Strasbourg, France